CLINICAL TRIAL: NCT02996630
Title: Abnormal Neurodevelopment Detection in Congenital Heart Disease: Predictive Methods Based on Prenatal and Postnatal Factors.
Brief Title: Assessing Neurodevelopment in Congenital Heart Disease.
Acronym: NEUROHEART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Sant Joan de Deu (Other); Hospital Universitario La Paz (Other); Hospital Universitario 12 de Octubre (Other); Hospital General Universitario Gregorio Marañon (Other); Fundacion Dexeus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR(AMI)317/2012
Record Dates: First submitted 2016-10-31; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-10

CONDITIONS: Congenital Heart Disease
Keywords: LVOTO; Fallot; Great Arteries Transposition
MeSH Terms: conditions — Heart Defects, Congenital; Transposition of Great Vessels | interventions — High-Energy Shock Waves; Magnetic Resonance Imaging; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy fetuses (Other): Pregnant patients carrying a healthy fetus. Interventions in this group will be: cord blood sample, sonography, Magnetic Resonance Imaging and bailey test.
  Interventions: Procedure: Sonography; Device: Magnetic Resonance Imaging; Other: Bailey Test; Procedure: cord blood sample
- Congenital Hearth Disease (Other): Pregnant patients carrying a fetus with a moderate-severe congenital heart disease Interventions in this group will be: cord blood sample, sonography, Magnetic Resonance Imaging, Surgical intervention, brain monitoring and bailey test.
  Interventions: Procedure: Sonography; Device: Magnetic Resonance Imaging; Other: Bailey Test; Procedure: Surgical intervention; Procedure: Brain monitoring; Procedure: cord blood sample

INTERVENTIONS:
Procedure: Sonography — Fetal Ultrasound exploration
Device: Magnetic Resonance Imaging — Fetal MRI for brain study
Other: Bailey Test — Neurodevelopment paediatric assessment test performed at 2 years of age.
Procedure: Surgical intervention — Congenital Heart Disease repair
  Arms: Congenital Hearth Disease
Procedure: Brain monitoring — EEG and continuous brain oximetry before surgery.
  Arms: Congenital Hearth Disease
Procedure: cord blood sample — Cord blood samples will be taken after birth in both groups.

SUMMARY:
Congenital heart disease (CHD) is the most prevalent congenital malformation affecting 1 in 100 newborns per year. Children with CHD are a known risk population for brain injury, with neurodevelopmental alterations shown over time in up to 50% of cases. No adequate description exists of the type of neurocognitive anomalies or risk factors associated with CHD, and consequently no prognostic markers that may allow identification of high-risk cases are available.

DETAILED DESCRIPTION:
The main objectives of this study are: 1. to describe the neurodevelopmental outcome of patients with CHD at 24 months of age; 2. identify the subgroup with poorer outcome; and 3. evaluate the utility of fetal and postnatal diagnostic techniques for early detection of patients at risk for altered neurological outcomes.

Seven Spanish referral centers for CHD included in the research network on maternal and child health currently participating in this prospective multicentric case-control coordinated study. Fetuses with CHD (transposition of great arteries, tetralogy of Fallot, hypoplastic left heart syndrome and septal defects) will be studied from 24 weeks of gestation to 2 years of age. Diagnostic tests will be repeated throughout the study in all patients, from the fetal period to 24 months of age, and will include: fetal cerebral hemodynamic Doppler assessment, functional echocardiography, brain MRI, regional cerebral oxymetry, electroencephalography and serum neurological and cardiac biomarkers analysis. Neurodevelopmental assessment will be made at 12 months of age using the ages and stages questionnaire (ASQ) and at 24 months of age with the Bayley-III test. From this data, statistical analysis will select the most useful as predictors of damage; to be then combined and create algorithms for predicting brain damage and poor neurodevelopment. Once description has been made, we will proceed to identify amongst our results, children with the poorest neurological outcome and remark possible common prenatal and early life markers in them as well as the CHD severity they present.

While advances in early diagnosis and postnatal management have increased survival in CHD children, worrying long-term outcomes, particularly neurodevelopmental disability, have emerged as a key prognostic factor in the counseling of these pregnancies. Evidence available does not allow clinicians to assess on neurological prognosis although has opened up the possibility of finding prenatal markers of brain damage. Even though, no prospective studies have been performed until now. We present a multicentric prospective study able to recruit enough fetal CHD affected pregnancies to obtain neurological prognostic tools.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancies
* Major Congenital Heart Disease
* Informed Consent Signed

Exclusion Criteria:

* Major extra-cardiac malformations
* Parental Refusal to participate
* Maternal Chronic Disease
* Multiple Pregnancies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Bailey-III test punctuation | 45 minutes
  Results in pediatric Bailey-III test scale

SECONDARY OUTCOMES:
Biparietal diameter (mm) | one day
  Biparietal diameter (mm) measured with MRI
Lateral sulcus depth | one day
  Lateral sulcus depth (mm) measured with MRI
Cerebral insula | one day
  Insula (mm) measured with MRI
Brain biometries | one day
  Calcarine sulcus depth (mm)
Cerebral cingulata sulcus | one day
  Cingulata sulcus depth (mm) measured with MRI
Corpus callosum | one day
  Corpus callosum (mm) measured with MRI
Cerebellum | one day
  Cerebellum vermis (mm) measured with MRI
Umbilical doppler | one day
  Umbilical artery pulsatility index
Middle cerebral artery doppler | one day
  Middle cerebral artery pulsatility index
Angiogenic PLGF (placental growth factor) | Two days
  Placental growth factor in maternal serum
Angiogenic s-FLt (soluble fms-like tyrosine kinase) | Two days
  Soluble fms-like tyrosine kinase factor in maternal serum

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Llurba, MD, PhD, Study Director — Hospital Universitari Vall d'Hebrón
Locations (1):
- Hospital Universitari Vall d'Hebrón, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Result] Bellinger DC, Jonas RA, Rappaport LA, Wypij D, Wernovsky G, Kuban KC, Barnes PD, Holmes GL, Hickey PR, Strand RD, et al. Developmental and neurologic status of children after heart surgery with hypothermic circulatory arrest or low-flow cardiopulmonary bypass. N Engl J Med. 1995 Mar 2;332(9):549-55. doi: 10.1056/NEJM199503023320901. PMID 7838188
- [Result] Limperopoulos C, Majnemer A, Shevell MI, Rosenblatt B, Rohlicek C, Tchervenkov C. Neurodevelopmental status of newborns and infants with congenital heart defects before and after open heart surgery. J Pediatr. 2000 Nov;137(5):638-45. doi: 10.1067/mpd.2000.109152. PMID 11060529
- [Result] Masoller N, Martinez JM, Gomez O, Bennasar M, Crispi F, Sanz-Cortes M, Egana-Ugrinovic G, Bartrons J, Puerto B, Gratacos E. Evidence of second-trimester changes in head biometry and brain perfusion in fetuses with congenital heart disease. Ultrasound Obstet Gynecol. 2014 Aug;44(2):182-7. doi: 10.1002/uog.13373. Epub 2014 Jul 8. PMID 24687311
- [Result] Ruiz A, Cruz-Lemini M, Masoller N, Sanz-Cortes M, Ferrer Q, Ribera I, Martinez JM, Crispi F, Arevalo S, Gomez O, Perez-Hoyos S, Carreras E, Gratacos E, Llurba E. Longitudinal changes in fetal biometry and cerebroplacental hemodynamics in fetuses with congenital heart disease. Ultrasound Obstet Gynecol. 2017 Mar;49(3):379-386. doi: 10.1002/uog.15970. PMID 27214694
- [Derived] Ribera I, Ruiz A, Sanchez O, Eixarch E, Antolin E, Gomez-Montes E, Perez-Cruz M, Cruz-Lemini M, Sanz-Cortes M, Arevalo S, Ferrer Q, Vazquez E, Vega L, Dolader P, Montoliu A, Boix H, Simoes RV, Masoller N, Sanchez-de-Toledo J, Comas M, Bartha JM, Galindo A, Martinez JM, Gomez-Roig L, Crispi F, Gomez O, Carreras E, Cabero L, Gratacos E, Llurba E. Multicenter prospective clinical study to evaluate children short-term neurodevelopmental outcome in congenital heart disease (children NEURO-HEART): study protocol. BMC Pediatr. 2019 Sep 10;19(1):326. doi: 10.1186/s12887-019-1689-y. PMID 31506079